CLINICAL TRIAL: NCT03744962
Title: A Compare of Microsatellite Instability in Circulatory DNA and Tumor Tissue of Endometrial Cancer
Brief Title: MSI in Circulatory DNA of Endometrial Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: EC-MSI
Record Dates: First submitted 2018-11-09; First posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Microsatellite Instability; Lynch Syndrome; Endometrial Cancer; Circulating Tumor Cell
MeSH Terms: conditions — Microsatellite Instability; Colorectal Neoplasms, Hereditary Nonpolyposis; Endometrial Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — An 8 ml peripheral venous blood, and 50 μL cancer tissue or tissue from from paraffin section will be collected from eligible patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to analyze the microsatellite instability (MSI) in the circulatory tumor DNA and in the tumor tissue in the patients diagnosed with uterine endometrial cancer. These data will be used for the study of "Cohort Study of Universal Screening for Lynch Syndrome in Chinese Patients of Endometrial Cancer" (NCT03291106, clinicaltrials.gov).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed primary endometrial cancer before any surgical or chemotherapy treatment
* Signed an approved informed consents
* Feasible for sampling

Exclusion Criteria:

* Not meeting all of the inclusion criteria

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients confirmed primary endometrial cancer before any surgical or chemotherapy treatment will be all included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-11-10 (Actual); Primary Completion 2020-12-23 (Estimated); Study Completion 2020-12-23 (Estimated)

PRIMARY OUTCOMES:
Frequency of microsatellite instability | Two years
  Frequencies of different status of microsatellite instability (high microsatellite instability or microsatellite-stable) in the circulatory tumor DNA and in the tumor tissue

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China